CLINICAL TRIAL: NCT06304493
Title: Postoperative Utilization of Incentive Spirometry With and Without Electronic Patient Reminders in the Post-Anesthesia Care Unit (PACU)
Brief Title: REMINDers for Incentive Spirometry in PACU (REMIND-IS in PACU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-2470
Record Dates: First submitted 2024-02-20; First posted 2024-03-12 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Atelectasis; Postoperative Hypoxemia; Postoperative Pneumonia; Postoperative Pulmonary Complications; Patient Adherence; Incentive Spirometry; Respiratory Therapy; Respiratory Insufficiency
Keywords: Incentive Spirometry; Postoperative Pulmonary Complications; Postoperative Standard-Of-Care; standard-of-care after surgery; Deep Breathing; Patient Reminders
MeSH Terms: conditions — Patient Compliance; Respiratory Insufficiency | interventions — Clinical Alarms

STUDY DESIGN:
Intervention Model Description: This is a pragmatic single-center cluster study of surgical patients receiving incentive spirometry devices during their PACU stay, with either automatic alarms "ON" or "OFF" in alternating weeks.
Who Masked: Outcomes Assessor
Masking Description: Outcome collection and data analysis will be performed by investigators blinded to the patient's cluster allocation (alarms "ON" or "OFF").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Alarm "ON" Cohort (Experimental): The "ON" cohort will receive the standard-of-care instructions for IS and information about the auditory and visual reminders. The "ON" cohort patients will receive audible and visual signals from the InSee monitor attached to their incentive spirometer every 20 minutes and upon successfully reaching certain achievements.
  Interventions: Device: Alarms
- Alarm "OFF" Cohort (Placebo Comparator): The "OFF" cohort will receive only the standard-of-care instructions for IS. The "OFF" patients will receive no signals from the InSee monitor attached to their incentive spirometer.
  Interventions: Device: Alarms

INTERVENTIONS:
Device: Alarms — The "ON" cohort patients will receive audible and visual signals from the InSee monitor attached to their incentive spirometer every 20 minutes and upon successfully reaching certain achievements.
  Other Names: Auditory and visual reminders

SUMMARY:
The purpose of this study is to determine if the frequency of use of incentive spirometry during the stay in the Post-Anesthesia Care Unit (PACU) increases with visual and auditory electronic reminders, as compared to not having those reminders.

DETAILED DESCRIPTION:
This is a pragmatic single-center alternating cluster study. We will enroll adult patients who require general anesthesia for surgery and receive an incentive spirometry device during their PACU stay. Automatic alarms to perform incentive spirometry will be set to either "ON" or "OFF" in alternating weeks. The hypothesis is that patients receiving automatic audible and visual alarms will have increased rates of adequate incentive spirometry breaths compared to patients receiving no alarms.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older;
* have undergone a surgical procedure at the University of Colorado Hospital under general anesthesia;
* have incentive spirometry ordered by their provider, or incentive spirometry must be part of the study site's standard-of-care which is implemented by hospital staff;
* not have severe hearing or impaired visual acuity deficiency, in that they cannot hear or see the audible and visual signal of the InSee monitor.

Exclusion Criteria:

* have a severe hearing or visual acuity impairment that prevents them from hearing or seeing the audible and visual signals of the InSee monitor;
* have the inability to perform incentive spirometry due to refusal, cognitive impairment, neuromuscular weakness, anatomical or any other reasons (e.g., tracheotomy, oral surgery, unable to hold incentive spirometry device);
* are a part of a vulnerable population (e.g., pregnant, minors, prisoners).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Rate of adequate IS breaths achieved in PACU | PACU stay (up to 3 hours)
  Rate of adequate incentive spirometry breaths achieved by patients per hour for up to 3 hours during the PACU stay

SECONDARY OUTCOMES:
Rate of IS breaths attempted in PACU | PACU stay (up to 3 hours)
  Rate of incentive spirometry breaths attempted by patients per hour for up to 3 hours during the PACU stay
Time to first adequate IS breath | PACU stay (up to 3 hours)
  The time it takes for the patient to achieve their first adequate IS breath, from the moment of being provided the IS device and instructions of use onward, during their PACU stay
Duration of postoperative O2 therapy | Hospital stay (up to first 3 postoperative days)
  The total postoperative length of oxygen therapy use from the time the patient arrives to PACU to the end of their O2 therapy
Presence of postoperative pulmonary complications | Hospital stay (up to first 3 postoperative days)
  The number of study participants developing any pulmonary complications (including pneumonia, need for non-invasive ventilation (CPAP/BiPAP or reintubation for any reason and any duration) during the first 3 postoperative days
Individual postoperative pulmonary complications | Hospital stay (up to first 3 postoperative days)
  The number of study participants developing each pulmonary complication (pneumonia, need for non-invasive ventilation (CPAP/BiPAP or reintubation for any reason and any duration) during the first 3 postoperative days
Need for ICU Admission after PACU | Hospital stay (up to first 3 postoperative days)
  The frequency of patients requiring ICU admission immediately after their PACU stay
PACU Length of Stay | PACU stay
  The length of stay in the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fernandez-Bustamante, MD, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- CU Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Shander A, Fleisher LA, Barie PS, Bigatello LM, Sladen RN, Watson CB. Clinical and economic burden of postoperative pulmonary complications: patient safety summit on definition, risk-reducing interventions, and preventive strategies. Crit Care Med. 2011 Sep;39(9):2163-72. doi: 10.1097/CCM.0b013e31821f0522. PMID 21572323
- [Background] Lawrence VA, Cornell JE, Smetana GW; American College of Physicians. Strategies to reduce postoperative pulmonary complications after noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):596-608. doi: 10.7326/0003-4819-144-8-200604180-00011. PMID 16618957
- [Background] Alwekhyan SA, Alshraideh JA, Yousef KM, Hayajneh F. Nurse-guided incentive spirometry use and postoperative pulmonary complications among cardiac surgery patients: A randomized controlled trial. Int J Nurs Pract. 2022 Apr;28(2):e13023. doi: 10.1111/ijn.13023. Epub 2021 Oct 22. PMID 34676618
- [Background] Bergin C, Speroni KG, Travis T, Bergin J, Sheridan MJ, Kelly K, Daniel MG. Effect of preoperative incentive spirometry patient education on patient outcomes in the knee and hip joint replacement population. J Perianesth Nurs. 2014 Feb;29(1):20-7. doi: 10.1016/j.jopan.2013.01.009. PMID 24461279
- [Background] Chang PC, Chen PH, Chang TH, Chen KH, Jhou HJ, Chou SH, Chang TW. Incentive spirometry is an effective strategy to improve the quality of postoperative care in patients. Asian J Surg. 2023 Sep;46(9):3397-3404. doi: 10.1016/j.asjsur.2022.11.030. Epub 2022 Nov 24. PMID 36437210
- [Background] Yanez-Brage I, Pita-Fernandez S, Juffe-Stein A, Martinez-Gonzalez U, Pertega-Diaz S, Mauleon-Garcia A. Respiratory physiotherapy and incidence of pulmonary complications in off-pump coronary artery bypass graft surgery: an observational follow-up study. BMC Pulm Med. 2009 Jul 28;9:36. doi: 10.1186/1471-2466-9-36. PMID 19638209
- [Background] Cassidy MR, Rosenkranz P, McCabe K, Rosen JE, McAneny D. I COUGH: reducing postoperative pulmonary complications with a multidisciplinary patient care program. JAMA Surg. 2013 Aug;148(8):740-5. doi: 10.1001/jamasurg.2013.358. PMID 23740240
- [Background] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Eltorai AEM, Szabo AL, Antoci V Jr, Ventetuolo CE, Elias JA, Daniels AH, Hess DR. Clinical Effectiveness of Incentive Spirometry for the Prevention of Postoperative Pulmonary Complications. Respir Care. 2018 Mar;63(3):347-352. doi: 10.4187/respcare.05679. Epub 2017 Dec 26. PMID 29279365
- [Background] Pantel H, Hwang J, Brams D, Schnelldorfer T, Nepomnayshy D. Effect of Incentive Spirometry on Postoperative Hypoxemia and Pulmonary Complications After Bariatric Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 May 1;152(5):422-428. doi: 10.1001/jamasurg.2016.4981. PMID 28097332
- [Background] Wesp JA, Duke MC, Farrell TM. Incentive Spirometry After Bariatric Surgery: Yes or No? JAMA Surg. 2017 May 1;152(5):428. doi: 10.1001/jamasurg.2016.4999. No abstract available. PMID 28097336
- [Background] Fernandez-Bustamante A, Schoen J, Vidal Melo MF. Incentive Spirometry After Bariatric Surgery: The Importance of Patient Compliance. JAMA Surg. 2017 Oct 1;152(10):984-985. doi: 10.1001/jamasurg.2017.1698. No abstract available. PMID 28636722
- [Background] Narayanan AL, Hamid SR, Supriyanto E. Evidence regarding patient compliance with incentive spirometry interventions after cardiac, thoracic and abdominal surgeries: A systematic literature review. Can J Respir Ther. 2016 Winter;52(1):17-26. PMID 26909010
- [Background] Eltorai AEM, Baird GL, Eltorai AS, Pangborn J, Antoci V Jr, Cullen HA, Paquette K, Connors K, Barbaria J, Smeals KJ, Agarwal S, Healey TT, Ventetuolo CE, Sellke FW, Daniels AH. Incentive Spirometry Adherence: A National Survey of Provider Perspectives. Respir Care. 2018 May;63(5):532-537. doi: 10.4187/respcare.05882. Epub 2018 Jan 23. PMID 29362219
- [Background] Zoremba M, Dette F, Gerlach L, Wolf U, Wulf H. Short-term respiratory physical therapy treatment in the PACU and influence on postoperative lung function in obese adults. Obes Surg. 2009 Oct;19(10):1346-54. doi: 10.1007/s11695-009-9922-7. Epub 2009 Jul 21. PMID 19626381